CLINICAL TRIAL: NCT05632900
Title: COMPARISON OF OUTCOMES OF BI-FLANGED METAL STENT ALONE VERSUS BI-FLANGED METAL STENT WITH CO-AXIAL PLASTIC STENT FOR DRAINAGE OF WALLED-OFF PANCREATIC NECROSIS
Brief Title: COMPARISON OF OUTCOMES OF BI-FLANGED METAL STENT ALONE VERSUS BI-FLANGED METAL STENT WITH CO-AXIAL PLASTIC STENT FOR DRAINAGE OF WALLED-OFF PANCREATIC NECROSIS - A PROSPECTIVE RANDOMISED CONTROLLED STUDY.
Acronym: BFMSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Doctor, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BFMSP -001
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: ENDOSCOPIC ULTRASONOGRAPHY

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAGI BI-FLANGED METAL STENT WITH CO-AXIAL PLASTIC STENT FOR DRAINAGE OF WOPN. (Experimental): Endoscopic ultrasound guided drainage -Nagi Bi Flanged metal stent--16mm diameter 2cm long with co Axial double pig tail stent used for drainage of walled of necrosis. Intra and post prodecural complications will be noted, a plane CT screening abdomen will be performed with in 48 to 72 hours to document the size of collection.
  Interventions: Procedure: Endoscopic ultrasound guided drainage of walled off pancreatic necrosis
- NAGI BI-FLANGED METAL STENT ALONE FOR DRAINAGE OF WOPN. (Active Comparator): Endoscopic ultrasound guided drainage -Nagi Bi Flanged metal stent--16mm diameter 2cm long used for drainage of walled of necrosis. Intra and post prodecural complications will be noted, a plane CT screening abdomen will be performed with in 48 to 72 hours to document the size of collection.
  Interventions: Procedure: Endoscopic ultrasound guided drainage of walled off pancreatic necrosis

INTERVENTIONS:
Procedure: Endoscopic ultrasound guided drainage of walled off pancreatic necrosis — It is Therapeutic procedure to treat walled off pancreatic necrosis.

SUMMARY:
Endoscopic ultrasound guided drainage of WON with metal stent is the mainstay of WON management.

But there are few complications related to BFMS , like bleeding due to vessel erosion, stent clogging , stent migration .

This study is to assess, whether placing an anchoring DPS through the BFMS will decrease adverse events or not.

There are only 2 retrospective studies till date ,comparing LAMS with coaxial stent vs LAMS alone.

one study showed no significant decrease in adverse events , one study showed decrease in adverse events when DPS with LAMS .

But there has been no prospective RCT to assess the utility of DPS to date

DETAILED DESCRIPTION:
Inclusion Criteria: -

1. Symptomatic Walled-off pancreatic necrosis (WON)
2. Eligible for EUS guided BFMS placement
3. Signed informed consent .
4. Age >18 Years

Exclusion Criteria: -

1. Types of pancreatic collections other than WON .
2. Drainage with stents other than BFMS
3. Previous attempts at drainage of WON
4. Coagulopathy (INR>1.5) or thrombocytopenia(plc <50000/cmm)- not correctable.
5. Pregnancy
6. Not willing to give informed consent

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic Walled-off pancreatic necrosis (WON)
2. Eligible for EUS guided BFMS placement
3. Signed informed consent .
4. Age >18 Years

Exclusion Criteria:

1. Types of pancreatic collections other than WON .
2. Drainage with stents other than BFMS
3. Previous attempts at drainage of WON
4. Coagulopathy (INR>1.5) or thrombocytopenia(plc <50000/cmm)- not correctable.
5. Pregnancy
6. Not willing to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-07-17 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Adverse evens rates associated with both the groups ( stent clogging and stent migration, bleeding). | 4 weeks
  To monitor the adverse events like bleeding, stent clogging and stent migration.

SECONDARY OUTCOMES:
re-intervention rates | 4 weeks
  Number of sessions of Direct Endoscopic necrosectomy and De clogging of stent
Technical success rate | 4 weeks
  Deployment of Stent
Clinical success rate | 4 weeks
  Resolution of symptoms Resolution of size of walled of necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Dr Gupta, MBBS MD DM, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Dr Rajesh Gupta, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No